CLINICAL TRIAL: NCT03786731
Title: A Transdiagnostic Sleep and Circadian Treatment for Major Depressive Disorder: A Randomised Controlled Trial
Brief Title: A Transdiagnostic Sleep and Circadian Treatment for Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: University of California, Berkeley (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY004
Record Dates: First submitted 2018-12-21; First posted 2018-12-26 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Major Depressive Disorder; Sleep Disturbance
Keywords: Major Depressive Disorder; Sleep; Transdiagnostic Sleep and Circadian Treatment
MeSH Terms: conditions — Depressive Disorder, Major; Parasomnias | interventions — Sleep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TranS-C Group (Experimental): Transdiagnostic Sleep and Circadian Treatment
  Interventions: Behavioral: Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C)
- CAU group (No Intervention): Care-As-Usual group

INTERVENTIONS:
Behavioral: Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C) — TranS-C integrates elements of evidence-based interventions, namely cognitive-behavioural therapy for insomnia, delayed sleep phase type, and interpersonal and social rhythm therapy.
  Arms: TranS-C Group

SUMMARY:
This study will examine the use of a transdiagnostic Sleep and Circadian Treatment (TranS-C) in treating Major Depressive Disorder (MDD) in Chinese adults. Sleep disturbance is highly comorbid with a range of psychological disorders, especially MDD. MDD is a major public health concern and a leading cause of disability worldwide. A shift in treatment perspectives, from a disorder-specific approach to a transdiagnostic approach, has been proposed. While the disorder-specific approach tends to understand and treat different mental disorders as independent psychological problems, the transdiagnostic approach aims to identify common clinical features (e.g. sleep disturbances) across a range of psychological disorders. The transdiagnostic approach would potentially facilitate timely dissemination of evidence-based psychological treatments and contribute to significant public health implications.

This study will be a randomized controlled trial on the efficacy of TranS-C for MDD. TranS-C integrates elements of evidence-based interventions, namely cognitive-behavioral therapy for insomnia, delayed sleep phase type, and interpersonal and social rhythm therapy. Prior to all study procedures, an online informed consent (with phone support) will be obtained from potential participants. Around 150 eligible participants will be randomly assigned to the TranS-C group or the care-as-usual control group (CAU group) in a ratio of 1:1. The randomization will be performed by an independent assessor using a computer-generated list of numbers. No deception is necessary. Participants in the TranS-C group will receive TranS-C once per week for 6 consecutive weeks respectively. The group treatment will be delivered by a clinical psychology trainee under the supervision of a clinical psychologist. The TranS-C group will complete a set of online/paper-and-pencil questionnaires before the treatment commences, 1-week, and 12-week after the treatment sessions are completed. The CAU group will complete the same set of online/paper-and-pencil questionnaires during the same periods.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong Citizen who is able to speak Cantonese and read Chinese;
2. Aged ≥ 18 years;
3. Presence of the DSM-IV diagnostic criteria of MDD based on Chinese-bilingual Structured Clinical Interview for DSM-IV (SCID);
4. Score on PHQ-9 is 10 or above;
5. More than 1 sleep or circadian problem according to the Sleep and Circadian Problem Checklist, including time needed to fall asleep more than 30 minutes for more than 3 nights per week, less than 6 hours of sleep per night or at least 9 hour of sleep per night per 24 hour period for at least 3 nights per week, variability in the sleep-wake schedule at least 2.78 hours within a week, and falling asleep after 2 am on at least 3 nights per week;
6. Adequate opportunity and circumstances for sleep to occur; and
7. Willing to give informed consent and comply with the trial protocol.

Exclusion Criteria:

1. Presence of other psychiatric disorders as defined by the DSM-IV diagnostic criteria using SCID;
2. Major medical or neurocognitive disorders that make participation infeasible;
3. Have suicidal ideation based on Beck Depression Inventory (BDI-II) Item 9 score ≥ 2;
4. Untreated sleep disorders based on SLEEP-50 (≥ 7 on narcolepsy; ≥ 15 on OSA; ≥ 7 on RLS/PLMD);
5. Past or current involvement in a psychological treatment programme for depression and/or sleep problems;
6. Shift work, pregnancy, work, family, or other commitments that interfere with regular night-time sleep patterns;
7. Hospitalization; and
8. A change in psychotropic drugs within 2 weeks before baseline assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Change in the Patient Health Questionnaire (PHQ-9) | Pre-treatment, 1-week post-treatment and 12-week post treatment]
  The PHQ-9, a 20-item questionnaire used for screening, diagnosing, monitoring and measuring the severity of depression, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day). PHQ-9 scores of 5, 10, 15, and 20 represents mild, moderate, moderately severe and severe depression

SECONDARY OUTCOMES:
Change in Hospital Anxiety and Depression Scale (HADS) | Pre-treatment, 1-week post-treatment and 12-week post treatment
  A 14-item self-rating scale that measures anxiety and depression in both hospital and community settings. It is divided into an Anxiety subscale (HADS-A) and a Depression subscale (HADS-D) both containing seven intermingled items. It is for screening purpose and not meant to be a diagnostic tool. HADS scores of 8-10, 11-14, and 15-21 represent mild, moderate, and severe anxiety and depression separately.
Change in Insomnia Severity Index (ISI) | Pre-treatment, 1-week post-treatment and 12-week post treatment
  A 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5-point Likert scale are obtained on the perceived severity of sleep-onset, sleep-maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem, and level of distress caused by the sleep problem. Total score categories: 0-7 is no clinically significant insomnia, 8-14 is subthreshold insomnia,15-21 is clinical insomnia (moderate severity), and 22-28 is clinical insomnia (severe)
Change in 7-Day Sleep Diary | Pre-treatment, 1-week post-treatment and 12-week post treatment
  The standardized sleep diary records sleep-onset latency (SOL; min), wake after sleep onset (WASO; min), total wake time (TWT; min), total sleep time (TST; min), time in bed (TIB; min); sleep efficiency (SE; calculated as TST/TIB * 100%), etc. Severity of sleep disturbances: sleep latency of time awake after sleep onset greater than 30 min; or last awakening occurring more than 30 min before desired time and before total sleep time reaches 6.5 hours; sleep efficiency is lower than 85%. Frequency: sleep difficulties present three or more nights per week.
Change in Multidimensional Fatigue Inventory (MFI) | Pre-treatment, 1-week post-treatment and 12-week post treatment
  A 20-item self-report instrument designed to measure fatigue. Ratings on a 5-point Likert scale are obtained on the dimensions of general fatigue, physical fatigue, mental fatigue, reduced motivation and reduced activity. Scores on each subscale range from 4 to 20, with higher scores indicating greater fatigue.
Change in Short Form (Six-Dimension) Health Survey - The Chinese (Hong Kong) Version (SF-6D) | Pre-treatment, 1-week post-treatment and 12-week post treatment
  A preference-based single index measure of health. A six-digit number represents each SF-6D health state, each digit denotes the level of one of six SF-6D dimensions: physical functioning, role limitation, social functioning, bodily pain, mental health, and vitality. The SF-6D index, scored from 0.0 (worst health state) to 1.0 (best health state)
Change in Sheehan Disability Scale (SDS) | Pre-treatment, 1-week post-treatment and 12-week post treatment
  A 5-item self-report tool for assessing functional impairment in work/school, social life, and family life. Representation of scores in terms of functional impairment: 0: not at all, 1-3: mildly, 4-6: moderately, 7-9: markedly, 10: extremely
Patient-Reported Outcomes Measurement Information System-Sleep Disturbance (PROMIS-SD) | Pre-treatment, 1-week post-treatment and 12-week post treatment
  PROMIS-SD item bank consists of 27 items and assesses perceptions of sleep quality, sleep depth, and restoration associated with sleep; perceived difficulties and concerns with getting to sleep or staying asleep; and perceptions of the adequacy of and satisfaction with sleep. PROMIS scores have a mean of 50 and standard deviation (SD) of 10 in a referent population. Scores 0.5 - 1.0 SD worse than the mean = mild symptoms/impairment. Scores 1.0 - 2.0 SD worse than the mean = moderate symptoms/impairment. Scores 2.0 SD or more worse than the mean = severe symptoms/impairment.
Patient-Reported Outcomes Measurement Information System-Sleep-Related Impairment (PROMIS-SRI) | Pre-treatment, 1-week post-treatment and 12-week post treatment
  The PROMISSRI item bank contains 16 items and assesses perceptions of alertness, sleepiness, and tiredness during usual waking hours, and the perceived functional impairments during wakefulness associated with sleep problems or impaired alertness. PROMIS scores have a mean of 50 and standard deviation (SD) of 10 in a referent population. Scores 0.5 - 1.0 SD worse than the mean = mild symptoms/impairment. Scores 1.0 - 2.0 SD worse than the mean = moderate symptoms/impairment. Scores 2.0 SD or more worse than the mean = severe symptoms/impairment

OTHER OUTCOMES:
Change in Credibility-Expectancy Questionnaire (CEQ) | Pre-treatment, 1-week post-treatment and 12-week post treatment
  The 6-item CEQ yielded ratings of treatment credibility, acceptability/satisfaction, and expectations for success. it measures how much the one believe that the therapy will help to improve one's lifestyle, functioning ranging from 1 to 9 with 1 representing the lowest value and the 9 representing the highest value. Two questions asking how much improvement in the functioning the one thinks and feels that it will occur ranging 0% to 100%. PROMIS scores have a mean of 50 and standard deviation (SD) of 10 in a referent population.
  Scores 0.5 - 1.0 SD worse than the mean = mild symptoms/impairment Scores 1.0 - 2.0 SD worse than the mean = moderate symptoms/impairment Scores 2.0 SD or more worse than the mean = severe symptoms/impairment

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Yau AY, Ng KY, Lau WY, Poon CY, Yeung WF, Chung KF, Chan CS, Harvey AG, Ho FY. A group-based transdiagnostic sleep and circadian treatment for major depressive disorder: A randomized controlled trial. J Consult Clin Psychol. 2024 Mar;92(3):135-149. doi: 10.1037/ccp0000869. Epub 2024 Jan 25. PMID 38271019